CLINICAL TRIAL: NCT01373983
Title: Evaluation of a Structured Algorithm for Intrathecal Bolus Doses of Ziconotide (Prialt®)- The Swedish Ziconotide Bolus Study
Brief Title: Intrathecal Bolus Doses of Ziconotide
Acronym: ZicBol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Emmanuel Backryd, Seniro Consultant in Pain management, University Hospital, Linkoeping
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: EudraCT 2010-018920-21
Record Dates: First submitted 2011-05-25; First posted 2011-06-15 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Peripheral Neuropathy
Keywords: Neuropathic pain; Intrathecal analgesia; Ziconotide; Bolus; trauma; central; severe; chronic
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia; Wounds and Injuries; Lymphoma, Follicular; Bronchiolitis Obliterans Syndrome | interventions — ziconotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ziconotide (Other)
  Interventions: Drug: Ziconotide

INTERVENTIONS:
Drug: Ziconotide — 1.25 or 2.5 mcg or 3.75 mcg i.t. according to an algorithm
  Other Names: Prialt

SUMMARY:
The purpose of this study is to evaluate if the effect of ziconotide can be tested by intrathecal bolus doses.

DETAILED DESCRIPTION:
The intrathecal route for administration of analgesia has been in use in clinical practice for the last 3 decades. It is recommended to trial the patient with intrathecal drug therapy prior to implanting an intrathecal drug delivery device. Trials can be performed using a single bolus injection or by a continuous intrathecal infusion administered through an external catheter. Ziconotide has been approved by EMA for the treatment of chronic severe pain in 2005. So far trials of ziconotide have largely been conducted using external catheters with the drug administered by intrathecal infusion over a number of weeks. Infusions trials have been shown to be expensive, associated with a risk of meningitis and inconvenient to both patient and physician. The option of conducting a trial of intrathecal ziconotide therapy by bolus injection remains unexplored.

This study aims to evaluate the efficacy and safety of a bolus dose of ziconotide (Prialt®) to evaluate the option of continuous administration of the drug via implanted pump in the event of a successful trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient, at least 18 years of age
* suffering from severe chronic (≥ 6 months) pain, who has failed on conventional pharmacological treatment
* only patients with peripheral neuropathic pain or central neuropathic pain, due to trauma or surgery, will be included
* Average usual VASPI last week ≥ 40 mm
* Patient capable of judgment, i.e. able to understand information regarding the drug, the mode of administration and evaluation of efficacy and side effects Signed informed consent

Exclusion Criteria:

* Limited life expectancy (investigator's judgement)
* Intrathecal chemotherapy
* Known or suspected intracranial hypertension
* Known liver or kidney disease, defined as ASAT, ALAT, Total Bilirubin, ALP or S- Creatinine > 1.2 x ULN
* Advanced cardio-pulmonary disease (investigator's judgment)
* Ongoing infection, whether systemically or locally in the lumbar area
* Coagulopathy (including medication with warfarin, clopidogrel and heparin)
* Allergy to ziconotide or any of the excipients in the ziconotide vial
* History of psychiatric disorders which in the investigator's opinion would put the patient at risk
* Pregnant or lactating woman.
* Menstruating women must use an effective contraceptive method (contraceptive pill or intrauterine spiral) during the trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale Pain Intensity, VASPI, 0-100 mm | VASPI before injection and then each hour after injection, for 6 hours.
  The average VASPI-score post-injection will be compared to the pre-injection value to yield a percentage pain reduction. Positive outcome is defined as a reduction of ≥30% in VASPI on two consecutive occasions at the same dosage without significant adverse events. All other cases will be considered as negative outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Bäckryd, MD, Principal Investigator — Pain and Rehabilitation Centre, University Hospital, Linköping, Sweden
Locations (1):
- Pain and Rehabilitation Centre, University Hospital, Linköping, Sweden

REFERENCES:
- [Derived] Jonsson M, Gerdle B, Ghafouri B, Backryd E. The inflammatory profile of cerebrospinal fluid, plasma, and saliva from patients with severe neuropathic pain and healthy controls-a pilot study. BMC Neurosci. 2021 Feb 1;22(1):6. doi: 10.1186/s12868-021-00608-5. PMID 33522900